CLINICAL TRIAL: NCT02212938
Title: Influence of a Standardised High Fat Breakfast on the Bioavailability of 10 mg BI 14332 CL Taken as Two Tablets of 5 mg q.d. in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-way Crossover Trial)
Brief Title: Influence of a Standardised High Fat Breakfast on the Bioavailability of BI 14332 CL in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1233.3
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BI 14332 CL fasted (Experimental)
  Interventions: Drug: BI 14332 CL
- BI 14332 CL fed (Experimental)
  Interventions: Drug: BI 14332 CL; Other: high fat breakfast

INTERVENTIONS:
Drug: BI 14332 CL
Other: high fat breakfast
  Arms: BI 14332 CL fed

SUMMARY:
To investigate the relative bioavailability of BI 14332 CL vs. BI 14332 CL after intake of a standardised high fat breakfast

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria:

Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests

* Age ≥21 and Age ≤65 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 192 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 192 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 192 hours after drug administration
AUCt1-t2 (partial area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | up to 192 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 192 hours after drug administration
λz (terminal rate constant in plasma) | up to 192 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 192 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 192 hours after drug administration
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | up to 192 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 192 hours after drug administration
Number of patients with adverse events | up to 23 days after last drug administration
Number of patients with clinically significant findings in vital signs (blood pressure, pulse rate) | up to 23 days after last drug administration
Number of patients with clinically significant findings in laboratory tests | up to 23 days after last drug administration
Number of patients with clinically significant findings in ECG | up to 23 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 23 days after last drug administration